CLINICAL TRIAL: NCT04783012
Title: Patient Removal of Urinary Catheters After Urogynecologic Surgery: A Randomized Non-Inferiority Trial
Brief Title: Patient Removal of Catheters After Urogynecologic Surgery
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-3376
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-03

CONDITIONS: Urinary Retention Postoperative; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home removal of catheter after surgery (Experimental): Patients randomized to home removal will be assigned to remove their catheters on postoperative day (POD) 2 (or if Th/F surgery, POD 4 or POD 3, respectively). They will be handed an instructional packed with visual, written and video instructions for catheter removal.
  Interventions: Procedure: Catheter removal
- Office removal of catheter after surgery (Active Comparator): Patients randomized to office removal will be assigned to return to the office on POD 2 (or if Th/F surgery, POD 4 or POD 3, respectively) for standard nurse visit with backfill, catheter removal and voiding trial in the office.
  Interventions: Procedure: Catheter removal

INTERVENTIONS:
Procedure: Catheter removal — Catheter management strategy after surgery

SUMMARY:
Management of postoperative urinary retention often requires the use of indwelling catheters. The purpose of this study is to see if patient removal of catheters at home is non-inferior to standard office removal.

DETAILED DESCRIPTION:
Voiding trials are a routine part of Urogynecologic surgery. Management of postoperative urinary retention often requires the use of indwelling catheters. However, patients often view the need for catheters as the worst part of their surgical experience, and follow-up voiding trials in the office utilize excess healthcare resources. Many Urology practices allow patient removal of catheters after procedures, though this has not been formally studied. The purpose of this study is to see if patient removal of catheters at home is non-inferior to standard office removal.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing prolapse or anti-incontinence surgery who fail their voiding trials prior to discharge
* 18+ years old

Exclusion Criteria:

* Non-English speaking
* Pregnant
* Elevated PVR (>150 mL) or dependent upon catheterization to void pre-operatively
* Urethral bulking injection surgery
* Intra-operative complication requiring prolonged catheterization
* Unable or unwilling to remove catheter at home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Risk of Urinary Retention in the Early Postoperative Period | 2-5 days postoperatively
  The percentage of patients who have urinary retention in the early postoperative period (failed voiding trial after discharge POD 2-5) will be measured.

SECONDARY OUTCOMES:
Number of nursing calls and office visits for urinary issues in the six week postoperative period | 6 week postoperative period
  Number of nursing calls and office visits for voiding issues (including catheter issues, voiding dysfunction and urinary retention) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Ijeoma Agu, MD, Principal Investigator — UNC Chapel Hill; Jennifer M Wu, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (2):
- United States (2):
  - UNC Hillsborough Hospital, Hillsborough, North Carolina
  - UNC Rex Hospital, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 to 36 months following publication
Access Criteria: Obtains approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Askew AL, Margulies SL, Agu I, LeCroy KM, Geller E, Wu JM. Patient Removal of Urinary Catheters After Urogynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2024 Feb 1;143(2):165-172. doi: 10.1097/AOG.0000000000005454. Epub 2023 Nov 14. PMID 37963385